CLINICAL TRIAL: NCT03081923
Title: An Open Label, Randomized, Phase 2 Study of the Anti-Programmed Death-Ligand 1 (PD-L1) Durvalumab, Alone or in Combination With Tremelimumab, in Patients With Advanced and Relapsed Germ Cell Tumors
Brief Title: Durvalumab Alone or With Tremelimumab in Refractory Germ Cell Tumors
Acronym: APACHE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: loss of accrual
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INT123-16
Record Dates: First submitted 2017-02-28; First posted 2017-03-16 (Actual); Last update posted 2021-05-14 (Actual); Status verified 2021-05

CONDITIONS: Germ Cell Tumor
Keywords: Immunotherapy; Durvalumab; Tremelimumab; Combination therapy; Testicular cancer
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Testicular Neoplasms | interventions — durvalumab; tremelimumab

STUDY DESIGN:
Intervention Model Description: Open-label, randomized, parallel arm, phase 2 trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Durvalumab (Experimental): Durvalumab, 1500 mg IV, q4 weeks, until disease progression or onset of unacceptable toxicity
  Interventions: Drug: Durvalumab
- Duralumab and Tremelimumab (Experimental): Durvalumab, 1500 mg IV, on day 1 and q4 weeks, until disease progression or onset of unacceptable toxicity Tremelimumab, 75 mg IV, both on day 1 and q4 weeks, until disease progression or onset of unacceptable toxicity
  Interventions: Drug: Durvalumab; Drug: Tremelimumab

INTERVENTIONS:
Drug: Durvalumab — anti-PD-L1 mono therapy
Drug: Tremelimumab — anti-CTLA4 drug Tremelimumab mono therapy
  Arms: Duralumab and Tremelimumab

SUMMARY:
Background:

The prognosis of pts who have failed multiple chemotherapy (CT) regimens is quite dismal. PD-L1 is frequently expressed by immunohistochemistry (IHC) in germ cell tumors (GCT). D is a monoclonal antibody (mAb) that inhibits the binding of PD-L1. T, an anti-CTLA4 mAb, is an immunomodulatory therapy. Combination immunotherapy has shown improved activity compared to monotherapy. The investigators aimed to investigate the activity of D, alone or in combination with T, in chemorefractory GCT.

Trial Design:

This is an open-label, randomized, 3-stage, phase 2 study. Pts who have failed ≥2 prior CT regimens (including high-dose CT) will be randomized to receive one of the following: D, 1.5 g via IV infusion q4w, for up to a total of 12 months (13 doses/cycles) alone or with T, 75 mg IV q4w, starting on week 0, for up to 4 months (4 doses/cycles). Serum tumor markers, computed tomography and fluorodeoxyglucose positron emission tomography (FDG-PET) scans will be repeated q8 weeks. The primary endpoint is the objective response-rate (ORR=complete response or partial response with normal markers). H0: ORR rate ≤10%, H1: ORR ≥25%, type I and II error rates at 10%.

In stage 1, 11 pts will be allocated in each arm. According to Gehan's rule, the trial will be terminated whenever no response will be observed. 29 additional pts will be added to each arm fulfilling stage 1 criteria. ORR in ≥7 pts will be required. In stage 3, pts from stage 1-2 of both arms will be retrospectively evaluated for Programmed cell Death Ligand-1(PD-L1) IHC. The Ventana PD-L1 IHC assay will be used. In case of negative findings at the end of stage 2, if the target benefit is likely to occur only in PD-L1+ pts, further study prosecution in accordance with an enrichment strategy will be undertaken.

In particular, predictive power (PP) will be calculated assuming expansion of PD-L1+ cohorts up to a maximum of 60 pts. Each arm will be categorized as not promising (PP<30%) or promising (PP ≥30%). The promising one will enter the stage 3. Should both arms be judged promising, the one yielding ≥20% PP advantage will be selected; monotherapy will be preferred otherwise. Details on the algorithm to be used for PD-L1 IHC in this study will be finalized (EudraCT number 2016-001688-35).

DETAILED DESCRIPTION:
This is an open-label, randomized, 3-stage, phase 2 study. Pts who have failed ≥2 prior CT regimens (including high-dose CT) will be randomized to receive one of the following: D, 1.5 g via IV infusion q4w, for up to a total of 12 months (13 doses/cycles) alone or with T, 75 mg IV q4w, starting on week 0, for up to 4 months (4 doses/cycles).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Male of female gender.
* Histological or clinical diagnosis of GCT.
* Availability of archival tumor samples for local assessment (by immunohistochemistry) of PD-L1 expression.
* Either gonadal or extragonadal tumor primary.
* Failure of ≥2 prior chemotherapy regimens for metastatic disease (1-2 cycles of cisplatin, etoposide and bleomycin (PEB) or 1 cycle carboplatin area under the curve (AUC) 7 given in the adjuvant setting for clinical stage I disease will not be counted as prior lines).
* Failure of high-dose chemotherapy will be allowed.
* Brain metastases: patients who present with brain metastases as the sole site of disease relapse/progression are not allowed to enter the study. Otherwise, patients with metastatic disease including brain metastases will be allowed provided that they have been irradiated, are stable from at least 4 weeks, and a wash-out period from steroids has occurred (28 days).
* Subjects must provide written informed consent.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Adequate end-organ system function tests.
* See the study full protocol for durvalumab-specific and tremelimumab requirements.

Exclusion Criteria:

* Prior exposure to immune-mediated therapy, including but not limited to, other anti-Cytotoxic T-Lymphocyte Antigen-4 (CTLA-4), anti-PD-1, anti-PD-L1, or anti-PD-L2 antibodies, including therapeutic anticancer vaccines.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Patients with Grade <2 neuropathy will be evaluated on a case-by-case basis after consultation with the Principal Investigator.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included after consultation with the Principal Investigator.
* Any concurrent chemotherapy, biologic, or hormonal therapy for cancer treatment.
* History of allogenic organ transplantation that requires use of immunosuppressive agents.
* Active or prior documented autoimmune or inflammatory disorders.
* Active infection including active tuberculosis, hepatitis B, hepatitis C, or human immunodeficiency virus (HIV).
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab or tremelimumab.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy or 180 days after the last dose of durvalumab + tremelimumab combination therapy.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2019-12-06 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Objective response-rate | 8 weeks
  Objective response-rate by computed tomography scan in accordance with the RECIST 1.1 criteria

SECONDARY OUTCOMES:
Overall survival | 6 months
  Number of subjects alive
Progression-free survival | 3 months
  Number of subjects alive and progression-free
Incidence of Adverse Events | 8 weeks
  Number of subjects developing side effects, graded according to the CTCAE v4.03

CONTACTS AND LOCATIONS:
Overall Officials: andrea necchi, MD, Principal Investigator — Fondazione IRCCS Istituto Nazionale tumori - Milano
Locations (1):
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Necchi A, Giannatempo P, Raggi D, Mariani L, Colecchia M, Fare E, Monopoli F, Calareso G, Ali SM, Ross JS, Chung JH, Salvioni R. An Open-label Randomized Phase 2 study of Durvalumab Alone or in Combination with Tremelimumab in Patients with Advanced Germ Cell Tumors (APACHE): Results from the First Planned Interim Analysis. Eur Urol. 2019 Jan;75(1):201-203. doi: 10.1016/j.eururo.2018.09.010. Epub 2018 Sep 19. No abstract available. PMID 30243800